CLINICAL TRIAL: NCT03802461
Title: Effectiveness of Fecal Flora Alteration for Eradication of Carbapenemase-producing Enterobacteriaceae Colonization Trial (EFFECT-CPE): a Multisite, Open-label, Randomized Controlled Feasibility Pilot Trial
Brief Title: Effectiveness of Fecal Flora Alteration for Eradication of Carbapenemase-producing Enterobacteriaceae Colonization
Acronym: EFFECT-CPE
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Temporarily on hold due to COVID-19 pandemic
Sponsor: Susy Hota (Other)
Collaborators: Sinai Health System, Ontario, Canada (Unknown); University of Toronto, Ontario, Canada (Unknown); The Toronto Invasive Bacterial Diseases Network, Ontario, Canada (Unknown); Public Health Ontario Laboratories, Ontario, Canada (Unknown)
Responsible Party: Sponsor-Investigator, Susy Hota, Medical Director, Infection Prevention and Control, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-5177
Record Dates: First submitted 2018-11-08; First posted 2019-01-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Infection
Keywords: Fecal Microbiota Transplantation; Gut Microbiome; Carbapenemase-producing Enterobacteriaceae (CPE)
MeSH Terms: conditions — Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Asymptomatic adult patients intestinally colonized with CPE will either randomized to receive fecal microbiota transplantation (intervention) or standard of care (no intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (FMT) (Active Comparator): Bowel lavage preparation followed by FMT administered by enema, given on 3 occasions. Fecal filtrate for FMT will be prepared from 50 g of healthy donor stool, homogenized, and diluted in 300 mL sterile normal saline.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)
- Standard of Care (No Intervention): Patients in this arm will not receive intervention and will be on standard of care .

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — Feces from healthy donor
  Arms: Fecal Microbiota Transplantation (FMT)

SUMMARY:
Carbapenemase-producing Enterobacteriaceae (CPE) are bacteria carried in the gastrointestinal tract that are resistant to carbapenems, antibiotics of last resort. CPE infections result in death in 25-50% of cases. Fecal microbiota transplantation (FMT) is the transfer of stool from a healthy donor to a recipient to alter the composition of gut microbes. Early studies support its use for eliminating CPE carriage but definitive studies are lacking. The investigators propose a feasibility pilot for a multicenter, non-blinded randomized trial comparing the effectiveness of FMT with no intervention (standard of care) in eliminating intestinal carriage of CPE. Forty patients with CPE will be randomly assigned to receive FMT by enema or no intervention. Feasibility will be demonstrated by the ability to recruit and retain 40 patients over 12 months, and to provide FMT made at a central site to at least one off-site hospital. The primary clinical endpoint for the full trial is CPE intestinal carriage 3 months after the intervention. Secondary endpoints include: CPE carriage at 1, 6 and 12 months; time to decolonization of CPE; safety; CPE infections over 12 months; and, intestinal carriage of other antibiotic-resistant organisms. Data on the clinical outcomes will be collected but not analyzed in this feasibility study.

DETAILED DESCRIPTION:
This is a multisite, open-label randomized controlled internal pilot trial designed to assess the feasibility of a larger trial aimed at determining the effectiveness of fecal microbiota transplantation (FMT) by enema in short and long term intestinal decolonization of carbapenemase-producing Enterobacteriaceae (CPE). Forty (40) asymptomatic adult patients intestinally colonized with CPE will be allocated in a 1:1 ratio to receive a bowel preparation followed by FMT by enema route, versus standard of care (no intervention). FMT will be provided by the University of Toronto Microbiota Therapeutics Outcomes Program (MTOP), using standardized operating procedures for recruiting and screening FMT donors, manufacturing FMT and administering FMT by enema. The feasibility outcomes are: successful randomization of 40 patients within 12 months, retention of >90% (36/40) of patients up to 6 months, and provision of FMT at a non-primary study site in at least one patient. Data on the clinical and exploratory outcomes will be collected but not analyzed in this pilot study. The primary clinical outcome is incidence of intestinal decolonization of CPE at 3 months. Secondary clinical outcomes include: time to decolonization of CPE; incidence of CPE clinical infections up to 12 months post-intervention; incidence of intestinal decolonization of CPE and other antibiotic-resistant organisms (extended spectrum beta-lactamase Enterobacteriaceae - ESBLs and vancomycin-resistant Enterococci - VRE) at 1, 3, 6 and 12 months post-intervention; and, safety profile. As an exploratory outcome, changes in fecal microbiome composition will be examined before and after intervention. This study leverages existing support, research infrastructures and expertise - including the Toronto Invasive Bacterial Diseases Network (TIBDN), Toronto Antimicrobial Resistance Research Network (TARRN), and the University of Toronto Microbiota Therapeutics Outcomes Program (MTOP) - to optimize feasibility regarding patient recruitment and FMT administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. ≥ 1 rectal swab, groin, stool, or urine specimen positive for a CPE within the past 1 month.

   • Presence of CPE will be confirmed at baseline through collection of pooled groin/rectal swab and urine specimen.
3. Women of childbearing age must be using at least one reliable form of birth control.
4. Must be able to provide informed consent.

Exclusion Criteria:

1. Active infection with CPE at the time of assessment.
2. Pregnancy, planned pregnancy or breastfeeding.
3. Current admission to intensive care unit.
4. Significantly immunocompromised patients .

   * neutropenia (ANC < 1)
   * ongoing use of systemic corticosteroids > 30 mg/day
   * ongoing use of biologic therapy
   * undergoing chemotherapy, received chemotherapy ≤ 30 days from baseline visit, or expected to undergo chemotherapy in the upcoming 12 months
   * active hematologic malignancy
   * solid organ transplant recipient
   * hematopoetic stem cell transplant recipient
   * HIV positive patients with cluster differentiation 4 (CD4) cell count < 350
5. Patients with ascites or receiving peritoneal dialysis.
6. History of inflammatory bowel disease (Crohn's or Ulcerative colitis).
7. Chronic diarrhea or active colitis for any reason.
8. Ileus or active gastrointestinal motility disorder at baseline.
9. History of total colectomy.
10. Severe, irreversible bleeding disorder.
11. History of anaphylactic or anaphylactoid allergic reaction to any foods.
12. Anticipated life expectancy less than 6 months.
13. Unable to tolerate enema.
14. Participant is not a Canadian citizen or permanent resident, and not expected to remain in Toronto region for 12 months.
15. Any reason in the view of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of intestinal colonization of patients with CPE 3 months after intervention. | 3 months
  Incidence of CPE colonization in FMT arm vs control arm at 3 months
Randomization rate in study | 12 months
  Completion of randomization of 40 study participants during the study period will be used to indicate feasibility of the study.
Proportion of patients retained in study for up to 6 months | 6 months
  A retention of 90% of patients up to 6 months in the study will be used to indicate feasibility.

SECONDARY OUTCOMES:
Incidence of CPE decolonization in FMT-treatment and non-treatment groups at 1, 6 and 12 months. | 1, 6, and 12 months
  As above
Time to CPE decolonization in FMT-treatment and non-treatment groups. | 1, 3, 6, and 12 months
  As above
Incidence of CPE clinical infection in FMT treatment and non-treatment groups over 12 months. | 1, 3, 6, and 12 months
  As above
Incidence of extended spectrum beta-lactamase organisms (ESBL) and vancomycin-resistant Enterococci (VRE) intestinal colonization at 0, 1, 3, 6 and 12 months in FMT treatment and non-treatment groups. | 1, 3, 6, and 12 months
  Changes in colonization status of other antimicrobial resistant organisms over the study period
Incidence of solicited and unsolicited adverse and serious adverse events in both groups | 3 months
  Participants will be asked to report adverse and serious adverse events will be throughout the study period and will be asked specifically about adverse events during study visits
Number of patients with all-cause mortality at 30 days post-randomization | 1 month
  As above

OTHER OUTCOMES:
Changes in composition and diversity of fecal bacterial phyla (as measured by 16s ribosomal ribonucleic acid sequencing) in both intervention groups | 12 months
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Susy S. Hota, MD MSc FRCPC, Principal Investigator — Infectious Diseases Physician, University Health Network; Susan M. Poutanen, MD MPH FRCPC, Principal Investigator — Microbiologist & Infectious Disease Physician, Sinai Health System
Locations (13):
- Canada (13):
  - William Osler Health System, Brampton, Ontario
  - Joseph Brant Hospital, Burlington, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - MacKenzie Health, Richmond Hill, Ontario
  - The Scarborough Hospital, Scarborough Village, Ontario
  - North York General Hospital, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Public Health Ontario Laboratories, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - St. Joseph Health Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No